CLINICAL TRIAL: NCT04282889
Title: Rotational Thromboelastometry (ROTEM) TRUE-NATEM Reference Value Validation in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 20D.086
Record Dates: First submitted 2020-02-18; First posted 2020-02-25 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Coagulation in Liver Transplantation
Keywords: ROTEM; Rotational Thromboelastometry; NATEM; TRUE-NATEM; Coagulation; liver transplantation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liver transplantation group: The study population will include 20 adults (age range of 18 - 75 years) who are undergoing liver transplantation. Inclusion criteria are patients undergoing liver transplantation with English as their native language.
  Exclusion criteria include patient's refusal, or on medical anticoagulation therapy. Informed consents will be obtained from the patients who agree to participate in this clinical study.
- Healthy volunteer: The control population will include 20 adult volunteers (age 18-65 years) who meet the in the American Society of Anesthesiologists (ASA) Physical Status (PS) Classes 1 criteria. Exclusion criteria will be refusal, volunteers on any medication or significant history of bleeding.

SUMMARY:
Background: Rotational thromboelastometry (ROTEM) has been used widely in liver transplantation for coagulation management. However, a TRUE-NATEM (TRUE-Non-Activated Rotational Thromboelastometry) reference value has never been established. A TRUE-NATEM value is of clinical significance since no coagulation activators or reagents will be added to the blood sample for analysis. Therefore, the result will reflect the true coagulation profile of the patient.

Methods: Non-citrated whole blood will be used for analysis. Blood will be drawn from the patient and transferred into a plastic reagent cup that has no reagent. Test will be performed within 4 minutes of blood draw to avoid activation of coagulation. Primary outcome measure will be clotting time (CT), clot formation time (CFT) and maximum clot firmness (MCF). The specific aims of the study are to establish a TRUE-NATEM reference value using Rotational Thromboelastometry (ROTEM®) in patients undergoing liver transplantation. Our hypothesis is that clotting time (CT), clot formation time (CFT) is prolonged and maximum clot firmness (MCF) decreased compared to healthy volunteers in patient undergoing liver transplantation due to synthetic coagulation factor deficiency.

DETAILED DESCRIPTION:
This study is a prospective cohort study establishing a TRUE-NATEM reference value using Rotational Thromboelastometry (ROTEM®) in patients undergoing liver transplantation.

The study population will include 20 adults (age range of 18 - 75 years) who are undergoing liver transplantation. Inclusion criteria are patients undergoing liver transplantation with English as their native language.

Exclusion criteria include patient's refusal, or on medical anticoagulation therapy. Informed consents will be obtained from the patients who agree to participate in this clinical study.

Currently, all patients undergoing liver transplantation will have hourly ROTEM analysis as standard of care. An additional TRUE-NATEM test will be performed after induction if anesthesia. 5 mL of whole blood will be obtained via a preexisting peripheral IV catheter or arterial line using a sterile technique. The blood will be transferred into a plastic reagent cup that has no additives. Test will be performed within 4 minutes of blood draw.3 All patients will undergo the standard anesthesia care and intraoperative coagulation monitoring and blood transfusion will be carried out using the standard practice guideline of the TJUH.

The control population will include 20 adult volunteers (age 18-65 years) who meet the in the American Society of Anesthesiologists (ASA) Physical Status (PS) Classes 1 criteria. Exclusion criteria will be refusal, volunteers on any medication or significant history of bleeding.

In the control group 5 mL of whole blood will be obtained after placing a peripheral IV catheter using a sterile technique. Blood draw from steel needle will be avoided because steel will activate coagulation. The blood will be transferred into a plastic reagent cup that has no additives. Test will be performed within 4 minutes of blood draw.

For each patient and control group four channels of ROTEM (TRUE-NATEM, NATEM, INTEM, EXTEM,) will be performed following the standard guideline at the Anesthesiology Coagulation Laboratory by a certified ROTEM specialists. Primary outcome measure will be clotting time (CT), clot formation time (CFT) and maximum clot firmness (MCF). The following demographic information will be collected; ASA physical status, age, height, weight, gender, home medication use, past medical history, and past surgical history.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are patients undergoing liver transplantation with English as their native language.

Exclusion Criteria:

* Exclusion criteria include patient's refusal, or on medical anticoagulation therapy. Informed consents will be obtained from the patients who agree to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include 20 adults (age range of 18 - 75 years) who are undergoing liver transplantation.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
clotting time (CT) | 1 year
  clotting time (CT) in seconds
clot formation time (CFT) | 1 year
  clot formation time (CFT) in seconds
maximum clot firmness (MCF) | 1 year
  maximum clot firmness (MCF) in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kang YG, Martin DJ, Marquez J, Lewis JH, Bontempo FA, Shaw BW Jr, Starzl TE, Winter PM. Intraoperative changes in blood coagulation and thrombelastographic monitoring in liver transplantation. Anesth Analg. 1985 Sep;64(9):888-96. PMID 3896028
- [Result] Durila M. Nonactivated thromboelastometry able to detect fibrinolysis in contrast to activated methods (EXTEM, INTEM) in a bleeding patient. Blood Coagul Fibrinolysis. 2016 Oct;27(7):828-830. doi: 10.1097/MBC.0000000000000479. PMID 26656899
- [Result] Meesters MI, Koch A, Kuiper G, Zacharowski K, Boer C. Instability of the non-activated rotational thromboelastometry assay (NATEM) in citrate stored blood. Thromb Res. 2015 Aug;136(2):481-3. doi: 10.1016/j.thromres.2015.05.026. Epub 2015 May 27. PMID 26044665